CLINICAL TRIAL: NCT03024723
Title: Comparison of Upper Airway Patency Using Continuous Positive Airway Pressure Ventilation Via a Nasal Mask With a Face Mask During Induction of Anesthesia on Obese Patients
Brief Title: Nasal Continuous Positive Airway Pressure and Airway Patency in Obese Patient
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yandong Jiang, Dr., Massachusetts General Hospital
Other Study IDs: 2013-P-000095/1
Record Dates: First submitted 2013-03-13; First posted 2017-01-19 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Obese
Keywords: Obese patient; nasal CPAP
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- FmCPAP: CPAP ventilation administered via face mask
  Interventions: Device: nasal mask CPAP

INTERVENTIONS:
Device: nasal mask CPAP — CPAP and ventilation administered via nasal mask
  Other Names: nCPAP

SUMMARY:
The mechanism of Upper airway obstruction (UAO) during anesthesia shares many similarities with the upper airway obstruction observed during obstructive sleep apnea (OSA). Nasal continuous positive airway pressure (nCPAP) via nasal mask (NM) can maintain the airway patent with near 100% success in patients with OSA. Obesity is a major risk factors for obstructive sleep apnea and obese patients have a higher prevalence of UAO during anesthesia. The investigators hypotheses that nCPAP should eliminate airway obstruction in obese patients under anesthesia. The investigators propose to test this hypothesis and determine the efficacy of nCPAP on maintaining airway patency in obese patients who require general anesthesia compared with CPAP administering face mask.

DETAILED DESCRIPTION:
Upper airway obstruction (UAO) is an unpredictable and frequently occurring complication during induction of general anesthesia. Since obese patients are more vulnerable to develop airway obstruction either during sleep1 or under anesthesia, and the segment of obese individuals in the entire population keep growing, difficult airway management under anesthesia becomes even more challenging than ever. The most serious event related to difficult airway management under anesthesia is "cannot intubate, cannot ventilate".

The mechanism of UAO during anesthesia has not been well understood. Obese patients are a high-risk group for perioperative airway catastrophe and prone to develop progressively narrower pharyngeal airways due to an increase of soft tissue volume surrounding the pharyngeal airway. The mechanism of UAO during anesthesia shares many similarities with the upper airway obstruction observed during obstructive sleep apnea (OSA). Nasal continuous positive airway pressure (nCPAP) via nasal mask (NM) can maintain the airway patent with near 100% success in patients with OSA. Obesity is a major risk factors for obstructive sleep apnea and obese patients have a higher prevalence of UAO during anesthesia. Therefore, the investigators hypotheses that nCPAP should eliminate airway obstruction in obese patients under anesthesia. The investigators propose to test this hypothesis and determine the efficacy of nCPAP on maintaining airway patency in obese patients who require general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

Body Mass Index:30 to 50 kg/ m2, Age: 18-65 years old ASA physical status classification: I-III Requiring general anesthesia for elective surgery

Exclusion Criteria:

1. Patients with major cardiovascular disease, respiratory disease, cerebral vascular disease or American Society of Anesthesiologists physical status class IV or greater.
2. Abnormal vital signs on the day of admission for surgery [heart rate (HR, >100 bpm or <40 bpm), blood pressure (BP, >180/100 mmHg or <90/60 mmHg), room air transcutaneous oxyhemoglobin saturation (SPO2) <96%] that are not correctable with his or her routine medication or commonly used pre-operative medication.
3. Having claustrophobia and not able to tolerate the mask.
4. Any person with an anticipated difficult airway or those with a history of difficult airway. This will include subjects who require or may require either a fiberoptic intubation or intubation while awake.
5. Gastric-esophageal reflex disease that is refractory to treatment or a full stomach.
6. The subject has been in bed for more than 24 hours.
7. Neurological symptoms associated with neck extension, a neurological deficit from a previous stroke or spinal cord injury, a recent stroke or transient ischemic attack (TIA) within 2 weeks.
8. Pregnant women and women less than one month post-partum. Ruling out pregnancy will be conducted by careful history and physical examination as performed routinely prior to surgery. If the history is believed to be unreliable, the patient will be excluded unless a pregnancy test is performed and the result of the test is negative.
9. Emergency cases and subjects who have not adhered to the ASA NPO (Nil Per Os) guidelines.

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult obese patient undergoing general anesthesia
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
expired tidal volume | 3 minutes
  This group of the subjects will start with nasal mask or face mask CPAP ventilation. The anesthesia care team does whatever they routinely do, including adjusting the patient's position (as to reverse Trendelenburg position), pre-oxygenation, pre-medication, as usual with intravenous anesthetics and analgesics. When the patient is apneic, CPAP ventilation will be initiated with pressure support mode at PIP 25 cmH2O, ventilation rate 10 BPM, PEEP 10 cmH2O and slope 1 second for 1 min. If ventilation is effective in one of the first three breaths, the ventilation will continue for 1 min. If effective ventilation cannot be produced in any of the first three breaths, the study will be terminated and routine care will be provided.

SECONDARY OUTCOMES:
expired tidal volume/Area under the Curve of the pressure trace | 3 minutes
  The area under the airway pressure curve (AUC) defined as the area from the baseline pressure to the peak pressure during inspiration was calculated for evaluating pressure applied during inspiration. The AUC is a reflection of the change in mean airway pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Yandong Jiang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States